CLINICAL TRIAL: NCT07030049
Title: Monocentric, Randomized Study, Comparing Articular Noise and Its Perception Between Two Different Types of Individualized Total Knee Arthroplasty
Brief Title: Comparing Articular Noise and Its Perception Between Two Different Types of Individualized Total Knee Arthroplasty
Acronym: ANIKA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Trenel (Other)
Collaborators: ProSurg (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 25.01072.000461; 2025-A00647-42 (Other: IDRCB national number)
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis; TKA
Keywords: osteoarthritis; TKA; articular noise
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: A randomised controlled single-blinded monocentre trial in a superiority framework with a 1:1 allocation ratio.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PS-group (Experimental): Individualized PS TKA
  Interventions: Device: Postero-stabilized total knee replacement for knee osteoarthritis
- CR-group (Active Comparator): Individualized CR TKA
  Interventions: Device: Cruciate-retaining total knee replacement for knee osteoarthritis

INTERVENTIONS:
Device: Postero-stabilized total knee replacement for knee osteoarthritis — Total knee arthroplasty in which the osteoarthritic knee is replaced with a postero-stabilized total knee replacement. The postero-stabilized TKA consists of a femoral component with a build-in cam mechanism and a tibial component with a post-mechanism.
  Arms: PS-group
Device: Cruciate-retaining total knee replacement for knee osteoarthritis — Total knee arthroplasty in which the osteoarthritic knee is replaced with a cruciate-retaining total knee replacement. The cruciate-retaining TKA consists of a femoral component and a tibial component that leaves the posterior cruciate ligament intact.
  Arms: CR-group

SUMMARY:
Knee osteoarthritis is a degenerative joint disorder leading to pain and limited movement. Total knee arthroplasty (TKA) has transformed the treatment of knee osteoarthritis, resulting in long-term outcomes that enhance the quality of life for patients. Some individuals report experiencing noise after undergoing TKA. However, there are few randomized controlled trials that assess postoperative noise following the procedure. Additionally, no research has been conducted on individualized TKA, which involves custom-made prostheses tailored to a patient's knee shape. This study aimed to compare the incidence of noise reported by patients who undergo a primary individualized TKA using either cruciate-retaining or posterior-stabilized designs.

DETAILED DESCRIPTION:
Articular noise is common after total knee arthroplasty (TKA), yet there is ongoing debate regarding its effect on postoperative outcomes, joint awareness and patient satisfaction. A comparative study on articular noise in 50 patients undergoing bilateral TKA using two different prosthesis designs reported that an ultra-congruent design generated less noise than a posterior-stabilized design (18% compared with 38%; p= 0.026), but there were no differences in patient preference, satisfaction, or Forgotten Joint Score (FJS) at two-year follow-up. A retrospective analysis of 160 robot-assisted and 320 conventional TKA revealed no difference in the prevalence of articular noise (40.7% vs 38.1%; p=0.647), but patients who complained of noise had lower FJS (45.5 vs 66.1; p<0.001) and lower Knee Injury and Osteoarthritis Score Joint Replacement (KOOS-JR) scores (72.0 vs 81.4; p<0.001) at one-year follow-up.

Recent advancements have shifted medicine from standardised approaches to personalised or precision medicine, tailoring treatments and decisions for individual patients based on their specific responses and risk factors. Individualized TKA adapts features to align with pre-arthritic anatomy and restore native movement, often utilising various tools. Recent studies on individualized TKA have demonstrated promising outcomes regarding personalised coronal alignment targets, correction of extra-articular deformities, intra-operative workflow, accommodation of the third compartment, and patient satisfaction rates.

This study will compare a posterior-stabilised (PS) and a cruciate-retaining (CR) individualized TKA implant. The PS implant is selected for patients with a damaged or a non-functional posterior cruciate ligament. In this case, the ligament is removed and substituted with a post-cam mechanism that aids femoral rollback during knee flexion and avoids anterior femoral subluxation. In contrast, the CR implant design can be selected for patients with an intact and functional posterior cruciate ligament. In this case, the ligament is retained, allowing it to guide femoral rollback and prevent anterior subluxation.

ELIGIBILITY:
Inclusion Criteria:

Adult patients:

* receiving elective primary TKA as a treatment for osteoarthritis
* with an intact and functional posterior cruciate ligament
* with no previous knee surgery, on the ipsi- or contra-lateral knee
* who signed the informed consent and are willing to comply with the protocol requirements based on the investigator's judgment.
* affiliated with a social security scheme
* with an ability to answer questionnaires and to communicate freely in French.

Exclusion Criteria:

Patients:

* that underwent previous knee surgery, except arthroscopic surgery, on their ipsilateral knee
* with coronal deformities >20°
* that are pregnant
* any contraindication mentioned in the instructions for use of the medical devices under investigation
* with protected status under articles L1121-6, LL121-8 and L1122-2 of the French Public Health Code
* with other significant disease or disorder which, in the opinion of the investigating surgeon, may put the participant at risk because of participation in the study, or may influence the result of the study
* who cannot comply with the protocol requirements based on the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Do you hear noise originating from your knee? | 2 years
  The surgeon will ask the blind participant whether they hear articular noise originating from their knee two years after TKA.

SECONDARY OUTCOMES:
Do you feel noise? | 1 & 2 years
  The surgeon will ask the blind participant whether they feel articular noise originating from their knee.
Is the noise a concern or causing discomfort? | 1 & 2 years
  The surgeon will ask the blind participant whether the articular noise originating from their knee is a concern or causing discomfort.
What kind of noise do you hear of feel? | 1 & 2 years
  The surgeon will ask the blind participant what kind articular noise originating from their knee (clunk, crepitus, grinding, clicking, other).
What part of the knee is involved? | 1 & 2 years
  The surgeon will ask the blind participant to identify which part of the knee is involved if they hear articular noise originating from their knee.
What is the impact of the noise on your quality of life, on a scale from 0 (none) to 10 (severe)? | 1 & 2 years
  The surgeon will ask the blind participant how their quality of life is affected by the articular noise originating from their knee.

OTHER OUTCOMES:
Forgotten Joint Score (FJS) | 1 & 2 years
  Patients will complete the 12-item forgotten joint score questionnaire. Scale: 0 (worst) to 100 (best)
Western Ontario et McMaster Universities Osteoarthritis Index (WOMAC) | 1 & 2 years
  Patients will complete the WOMAC questionnaire (3 domains: pain, stiffness and physical function). Scale: 0 (best) to 96 (worst).
Range of motion. | 1 & 2 years
  Clinical evaluation of knee mobility, using measurements of maximum flexion, flexion contracture (FC) and total range of motion (RoM) pre- and post-operatively.
Pain assessment using the numeric scale | 1 & 2 years
  Pain assessment on a numeric scale from 0 to 10.
Patient satisfaction | 1 & 2 years
  Patient satisfaction assessed using 5-point Likert scale (very satisfied, satisfied, neutral, dissatisfied, very dissatisfied).
Patient quality of life (QoL) | 1 & 2 years
  Patient QoL using the EQ-5D-5L questionnaire. Scale: -0.59 (worst) to 1.0 (best)
Analysis of adverse events | 0 to 2 years
  Analysis of adverse events: incidence, severity, and relationship to the medical device.

IPD SHARING:
Plan to Share IPD: No
It goes against GDPR and other EU regulations